CLINICAL TRIAL: NCT06552104
Title: The Effects of Acupressure Applied to the Primiparous During Episiotomy Repair on Pain and Anxiety Levels
Brief Title: The Effects of Acupressure Applied to the Primiparous During Episiotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esra SABANCI BARANSEL (Other)
Responsible Party: Sponsor-Investigator, Esra SABANCI BARANSEL, Assistant professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/ 4576
Record Dates: First submitted 2024-08-01; First posted 2024-08-13 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Episiotomy Wound; Pain; Anxiety
Keywords: Acupressure; episiotomy; primiparous
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACUPRESSURE (Experimental): In the study, acupressure was applied to the LI4 and HT7 points of the women for approximately 8-11 minutes during the episiotomy repair by BI, one of the researchers who has an acupressure application certificate. The researcher received training and certification in acupressure techniques before starting the intervention.During the episiotomy repair, acupressure was applied by the researcher twice in total. The first acupressure application was started with the first episiotomy suture being placed during the episiotomy repair (with the start of the internal perineal suturing). The second acupressure application was started with the end of the internal perineal suture and the first episiotomy suture of the skin suture. Each application was applied for approximately 4-6 minutes.
  Interventions: Behavioral: ACUPRESSURE APPLI ACUPRESSURE APPLICATION
- Control group (No Intervention): control groups Control group standard care group

INTERVENTIONS:
Behavioral: ACUPRESSURE APPLI ACUPRESSURE APPLICATION — Pre-test data were collected from participants who met the inclusion criteria and volunteered to participate in the study by researcher BI in the LDP rooms during the latency period of labor. Post-test data were obtained by the same researcher 16 hours after the cesarean section. Data were obtained using the Personal Information Form, Episiotomy Evaluation Form (EEF), Visual Analog Scale (VAS), and Spielberger Manual for State-Trait Anxiety Inventory (STAI).
  Arms: ACUPRESSURE

SUMMARY:
This study was conducted to determine the effects of acupressure applied during episiotomy repair on pain and anxiety levels of the primiparous.

The study was conducted as a randomized controlled trial with 126 pregnant women (63 women in the acupressure group and 63 women in the control) who applied to a maternity hospital between June and December 2023. Acupressure was applied to the acupressure group twice (during internal suturing and skin suturing) by the researcher during the episiotomy repair. Visual Analog Scale (VAS) was used a total of four times, before and after the intervention, to assess the pain scores of the participants, while the Spielberger Manual for State-Trait Anxiety Inventory (STAI) was used after the second intervention to determine the anxiety levels of the participants.

DETAILED DESCRIPTION:
Introduction: This study was conducted to determine the effects of acupressure applied during episiotomy repair on pain and anxiety levels of the primiparous.

Methods: The study was conducted as a randomized controlled trial with 126 pregnant women (63 women in the acupressure group and 63 women in the control) who applied to a maternity hospital between June and December 2023. Acupressure was applied to the acupressure group twice (during internal suturing and skin suturing) by the researcher during the episiotomy repair. Visual Analog Scale (VAS) was used a total of four times, before and after the intervention, to assess the pain scores of the participants, while the Spielberger Manual for State-Trait Anxiety Inventory (STAI) was used after the second intervention to determine the anxiety levels of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 or older,
* having a single healthy newborn,
* Giving spontaneous birth through a medio-lateral episiotomy incision,
* No signs of infection such as vaginal redness or swelling,
* Women with full and healthy tissue integrity in the area where acupressure will be applied.

Exclusion Criteria:

* The need to use unusual lidocaine during episiotomy repair (lidocaine 2% higher than 5 ml),
* having any postpartum complications (such as bleeding, hypertension).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Episiotomy is performed on women who have given birth.
Enrollment: 126 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
VAS | Change inbreastfeeding self-efficacy levels at 6 weeks change in pain after acupressure
  The VAS was used to assess the pain severity of the incision site. The VAS is a scale created in the range of 0-100 mm. According to the scale, a score of 0 mm indicates that the pain is not severe at all, and a score of 100 mm indicates that the pain is extremely severe

SECONDARY OUTCOMES:
STAI | Change inbreastfeeding self-efficacy levels at 6 weeks change in anxiety after acupressure
  STAI was developed by Spielberger et al. (1970) to measure state and trait anxiety levels, and its adaptation, validity, and reliability study was conducted by Öner and Le Compte (1983) for the Turkish society. The STAI is a 20-item inventory, and a high score indicates that the individual has a high level of anxiety, while a low score indicates that the anxiety level is low. The lowest score that can be obtained from the scale is 20, and the highest score is 80. This scale, which is a 4-point Likert-type scale, is graded as Not at All, A Little, A Lot, and Extremely.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Sabancı baransel, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No